CLINICAL TRIAL: NCT03558880
Title: Ultrasound Guided Bilateral Erector Spinae Plane Block Versus Tumescent Anesthesia in Reduction Mammoplasty
Brief Title: Ultrasound Guided Bilateral Erector Spinae Plane Block Versus Tumescent Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/11-20
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Breast Hypertrophy; Pain, Postoperative
MeSH Terms: conditions — Gigantomastia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Before the general anesthesia Erector Spinae Plane Block was performed.
  Interventions: Procedure: Erector Spinae Plane Block
- Tumescent Anesthesia (Active Comparator): After the general anesthesia was given, 1 mL of 0.1% adrenaline (1/1000) and as 20 mL of 0.5% bupivacaine solution of tumescent in a total of 1000 mL Ringer's lactate applied by the surgeon applied equally to both breasts
  Interventions: Procedure: Tumescent Anesthesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block was performed
  Arms: Erector Spinae Plane Block
Procedure: Tumescent Anesthesia — Tumescent Anesthesia was applied
  Arms: Tumescent Anesthesia

SUMMARY:
In breast reduction surgery, pain control is usually performed with tumescent anesthesia, thoracic epidural anesthesia, intercostal nerve blocks and paravertebral block applications. Tumescent anesthesia is also preferred by plastic surgeons because of the varying risk of thoracic epidural anesthesia and paravertebral block applications.

After the Erector spinae block was first described by Forero in 2016, it was reported to have been applied in many cases, including breast surgery.

It is considered to be a safer block because of the presence of paravertebral block-like activity and the location where the needle is guided away from the pleura. The investigators aimed to compare postoperative analgesia consumption, pain scores and patient satisfaction of erector spine block with tumescent anesthesia in patients who underwent reduction mammoplasty operation under general anesthesia in this double-blind prospective randomized study.

DETAILED DESCRIPTION:
Patients aged 18-65 years undergoing bilateral reduction mammoplasty. Patients were randomly divided into two groups with closed envelope to perform tumescent anesthesia and erector spinae block.

All patients were premedicated with oral midazolam 0.5 mg/ kg preoperatively. All patients received standard general anesthesia protocol as induction with 2-3 mg/kg iv propofol and 1-1.5 mcg/kg fentanyl and 0.6 mg/kg iv rocuronium. Endotracheal intubations were performed 7.0 or 7.5 endotracheal tubes with the patient in a supine position. Anesthesia maintenance was with sevoflurane 0.5/kg/mg remifentanil infusion and in a 50% O2 -50% air mixture. Standard monitoring of the patients included of heart rate, invasive systolic, diastolic and mean blood pressure and peripheral oxygen saturation and the operating times were recorded.

At approximately 30 minutes before the end of surgery, 8mg dexketoprofen IV was administered to all patients. At the end of the operation, all the patients were performed with iv PCA(Patient Controlled Analgesia).

Demographic data such as age, weight, and height of the patients were recorded. After patients informed about pain score NRS (Numeric Pain Rating Scale) and patient satisfaction score ( one to ten) recorded by the nurse of PACU and ward.

ELIGIBILITY:
Inclusion Criteria:

The American Society of Anesthesiologists physical status classification I-III undergoing reduction mammoplasty

Exclusion Criteria:

History of allergic reactions to local anesthetics Rash or infection at the injection site Anatomical abnormality Bleeding diatheses Coagulopathy liver diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Use of analgesic consumptions | 24 hour
  Total tramadol consumptions with patient controlled device

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 30 minute, 1,2,4,6,12,24 hour
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Gözen Öksüz, M.D., Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016